CLINICAL TRIAL: NCT05239117
Title: Open, Non-comparative, Multicentre Clinical Investigation to Evaluate the Performance and Safety of the Medical Device Plenhyage® (Polymerised Polynucleotides Dermal Filler) in the Treatment of Dermal Tissue Defects
Brief Title: Evaluating the Performance and Safety of the Medical Device Plenhyage® in the Treatment of Dermal Tissue Defects
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: I.R.A. Istituto Ricerche Applicate S.p.A. (Network)
Collaborators: Opera CRO, a TIGERMED Group Company (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: OPIRA/0521/MD
Record Dates: First submitted 2022-01-17; First posted 2022-02-14 (Actual); Last update posted 2022-10-25 (Actual); Status verified 2022-04

CONDITIONS: Cicatrix; Lipodystrophy; Plaque
MeSH Terms: conditions — Cicatrix; Lipodystrophy; Plaque, Amyloid

STUDY DESIGN:
Intervention Model Description: This is a multi-center, open-label, non-randomized clinical investigation
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Plenhyage Thin (Experimental): Sixteen patients will be administered Plenhyage® Thin for the treatment of minor -sized dermal tissue defects (scars, atrophic scars, depressed plaques, and lipodystrophy defects).
  Interventions: Device: Plenhyage
- Plenhyage Medium (Experimental): Sixteen patients will be administered Plenhyage® Medium for the treatment of medium-sized dermal tissue defects (scars, atrophic scars, depressed plaques, and lipodystrophy defects).
  Interventions: Device: Plenhyage
- Plenhyage Strong (Experimental): Sixteen patients will be administered Plenhyage® Strong for the treatment of major-sized dermal tissue defects (scars, atrophic scars, depressed plaques, and lipodystrophy defects).
  Interventions: Device: Plenhyage

INTERVENTIONS:
Device: Plenhyage — Plenhyage® is an elastic, sterile, injectable, non-pyrogenic, re-absorbable gel made with polymerised polynucleotides (PDRN) of animal origin (fish). Due to its hydrophilic and polyanionic nature, PDRN binds water molecules, thereby filling intradermal spaces and making tissues firmer and more hydrated.
  The polynucleotide chain binds water molecules, has an anti-free radical action, and serves as a scavenger of hydroxyl radicals (OH), which accumulate under stress or due to foreign agents, such as UV radiation. Its hydration and anti-free radical activity help create the optimal environment for fibroblast growth, thereby restoring tissue elasticity.
  Plenhyage® is a colourless gel contained in a pre-filled, graduated, disposable, and sterile syringe with a Luer Lok adapter.

SUMMARY:
The Research Question of the present study is the following: in a population of men and women presenting dermal tissue defects (scars, atrophic scars, depressed plaques, and lipodystrophy defects) will Plenhyage® significantly improve the appearance of treated areas, results observed after 4, 8 and 12 weeks?

DETAILED DESCRIPTION:
Plenhyage® is a different type of dermal filler, an innovative course of polynucleotides to restore skin damage. The polynucleotide chain attracts water molecules, protecting against free radicals, acting as an absorber of hydroxyl radicals OH, which accumulate from stress, cell damage and UV rays. It also guarantees moisturising action and protection against free radicals. Nucleotides, natural fractions of DNA and RNA, are components of Plenhyage® with an antioxidant, protective effect. These characteristics allow Plenhyage® to be used as a temporary filler for subcutaneous areas to correct small defects in the dermal tissue due to lipodystrophies or the presence of fibrotic tissues as scars, caused by pathologies or trauma.

ELIGIBILITY:
Inclusion Criteria:

1. Men or women with age ≥ 18 and ≤ 65 years.
2. Patients presenting dermal tissue defects (scars, atrophic scars, depressed plaques, and lipodystrophy defects), seeking tissue augmentation treatment and willing to receive Polymerized Polynucleotides Filler.
3. Patients who agree to discontinue any other dermatological treatment and procedures during the study.
4. Patients willing to provide signed informed consent to clinical investigation participation.
5. Patients able to communicate adequately with the Investigator and to comply with the requirements for the entire study.

Exclusion Criteria:

1. Use of aspirin and antiplatelet agents a week prior to treatment.
2. Patients with history of allergy or hypersensitivity to polymerised polynucleotides or to other ingredients of the dermal filler or hypersensitivity skin reaction to the investigational device based on intradermal test results at visit 1.
3. Patients with any dermal systemic pathologies, such as systemic lupus erythematosus, psoriasis, scleroderma etc..
4. Patients presenting bleeding disorders in the past or present.
5. Patients taking or having indications for anticoagulant therapy.
6. Use of concomitant treatments or procedures aimed to improve skin appearance over the last six months before the clinical investigation enrolment, such as chemical peeling, dermabrasion, laser resurfacing.
7. Patients suffering from infectious diseases including herpes simplex virus infection, active hepatitis or human immunodeficiency virus.
8. Patients suffering from active eczema, acne and keloids.
9. Patients with any cutaneous manifested infection, disease or alteration.
10. Patients at risk in term of precautions, warnings and contra-indications referred in the package insert of the clinical investigation device.
11. Patients with any facial aesthetic surgery in the preceding 12 months before the clinical investigation enrolment
12. Patients with any active irritation or inflammation in the target areas of injection.
13. Patients who received botulinum toxin A injections in the face in the preceding 6 months.
14. Patients unlikely to cooperate in the clinical investigation or to comply with the treatment or with the clinical investigation visits.
15. Pregnant woman, lactating woman, and man or woman of childbearing potential who is planning a pregnancy or is unwilling to use appropriate methods of contraception* during the study.

    *Methods of contraception: hormonal contraceptive, intrauterine device or intrauterine system, double barrier method (condom with spermicide/diaphragm or cervical cap with spermicide), surgical sterilization (vasectomy, tubal ligation, etc.).
16. Patients with illness, or other medical condition that, in the opinion of the Investigator, would compromise participation or be likely to lead to hospitalization during the study.
17. Participation in an interventional clinical study or administration of any investigational agents in the previous 30 days.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2022-03-30 (Actual); Primary Completion 2022-12-30 (Estimated); Study Completion 2022-12-30 (Estimated)

PRIMARY OUTCOMES:
POSAS score assessed by Investigator and patient | 8 weeks
  To evaluate the overall performance of the medical dermal filler Plenhyage® in treating dermal tissue defects (scars, atrophic scars, depressed plaques, and lipodystrophy defects) in terms of change in Patient and Observer Scar Assessment Scale (POSAS) score [Draaijers, 2004; van de Kar, 2005], assessed by Investigators and patients at 8 weeks ( 56 days) after the initiation of treatment, compared to Visit 1 (day 0)
POSAS score assessed by Investigator and patient | 4 weeks
  To evaluate the overall performance of the medical dermal filler Plenhyage® in treating dermal tissue defects (scars, atrophic scars, depressed plaques, and lipodystrophy defects) in terms of change in Patient and Observer Scar Assessment Scale (POSAS) score [Draaijers, 2004; van de Kar, 2005], assessed by Investigators and patients at 4 (28 days) after the initiation of treatment, compared to Visit 1 (day 0)
POSAS score assessed by Investigator and patient | 12 weeks
  To evaluate the overall performance of the medical dermal filler Plenhyage® in treating dermal tissue defects (scars, atrophic scars, depressed plaques, and lipodystrophy defects) in terms of change in Patient and Observer Scar Assessment Scale (POSAS) score [Draaijers, 2004; van de Kar, 2005], assessed by Investigators and patients at 12 weeks (84 days) after the initiation of treatment, compared to Visit 1 (day 0)
Investigator Global Assessment of Performance (IGAP) | 12 weeks
  To evaluate the global performance of product assessed by Investigator through photos taken at each visit (IGAP), at week 12 (day 84), compared to Visit 1 (day 0)
Adverse Event incidence | 12 weeks
  To evaluate the safety of the device through Adverse Event incidence assessed by Investigators at all visits and reported according to the current legislation
Serious Adverse Event incidence | 12 weeks
  To evaluate the safety of the device through Serious Adverse Event incidence assessed by Investigators at all visits and reported according to the current legislation
Adverse Device Event incidence | 12 weeks
  To evaluate the safety of the device through Adverse Device Event incidence assessed by Investigators at all visits and reported according to the current legislation
Serious Adverse Device Event incidence | 12 weeks
  To evaluate the safety of the device through Serious Adverse Device Event incidence assessed by Investigators at all visits and reported according to the current legislation
Device deficiency incidence | 12 weeks
  To evaluate the safety of the device through Device deficiency incidence assessed by Investigators at all visits and reported according to the current legislation

SECONDARY OUTCOMES:
Global Aesthetic Improvement Scale evaluated by the patient (GAIS) | 12 weeks
  To evaluate general appearance after treatment assessed by the patient at 4, 8 and 12 weeks (28, 56 and 84 days) using the Global Aesthetic Improvement Scale (GAIS) [Kim, 2016], [Kopera, 2015 - 2018], [McCall-Perez, 2011], [Savoia, 2015]. The scale evaluates the appearance from 1 (very much improved) to 5 (worse than original condition) .
Treatment satisfaction assessment by the patient | 12 weeks
  To assess the patient satisfaction at 4, 8 and 12 weeks (28, 56 and 84 days), providing their degree of satisfaction with the treatment on a four-point scale (very satisfied, satisfied, moderately satisfied, or not satisfied)
Investigator Global Assessment of Safety (IGAS) | 12 weeks
  To evaluate the global safety of product assessed by Investigator (IGAS), at week 12 (day 84), compared to Visit 1 (day 0), providing the safety on a four point scale from 4 meaning poor safety to 1 meaning very good safety.
Patient Global Assessment of Safety (PGAS). | 12 weeks
  To evaluate the global safety of product assessed by the patient (PGAS), at week 12 (day 84), compared to Visit 1 (day 0), providing the safety on a four point scale from 4 meaning poor safety to 1 meaning very good safety.

CONTACTS AND LOCATIONS:
Overall Officials: Mihaela Fratila, Principal Investigator — SCM Dr. Rosu
Locations (1):
- SCM Dr. Rosu, Timișoara, Timiș County, Romania

REFERENCES:
- [Background] Ascher B, Bayerl C, Brun P, Kestemont P, Rzany B, Poncet M, Guennoun M, Podda M. Efficacy and safety of a new hyaluronic acid dermal filler in the treatment of severe nasolabial lines - 6-month interim results of a randomized, evaluator-blinded, intra-individual comparison study. J Cosmet Dermatol. 2011 Jun;10(2):94-8. doi: 10.1111/j.1473-2165.2011.00550.x. PMID 21649813
- [Background] Barnes LA, Marshall CD, Leavitt T, Hu MS, Moore AL, Gonzalez JG, Longaker MT, Gurtner GC. Mechanical Forces in Cutaneous Wound Healing: Emerging Therapies to Minimize Scar Formation. Adv Wound Care (New Rochelle). 2018 Feb 1;7(2):47-56. doi: 10.1089/wound.2016.0709. PMID 29392093
- [Background] Beasley KL, Weiss MA, Weiss RA. Hyaluronic acid fillers: a comprehensive review. Facial Plast Surg. 2009 May;25(2):86-94. doi: 10.1055/s-0029-1220647. Epub 2009 May 4. PMID 19415575
- [Background] Bhatt A. Protocol deviation and violation. Perspect Clin Res. 2012 Jul;3(3):117. doi: 10.4103/2229-3485.100663. No abstract available. PMID 23125964
- [Background] Bogdan Allemann I, Baumann L. Hyaluronic acid gel (Juvederm) preparations in the treatment of facial wrinkles and folds. Clin Interv Aging. 2008;3(4):629-34. doi: 10.2147/cia.s3118. PMID 19281055
- [Background] Brandt FS, Cazzaniga A. Hyaluronic acid gel fillers in the management of facial aging. Clin Interv Aging. 2008;3(1):153-9. doi: 10.2147/cia.s2135. PMID 18488885
- [Background] Bukhari SNA, Roswandi NL, Waqas M, Habib H, Hussain F, Khan S, Sohail M, Ramli NA, Thu HE, Hussain Z. Hyaluronic acid, a promising skin rejuvenating biomedicine: A review of recent updates and pre-clinical and clinical investigations on cosmetic and nutricosmetic effects. Int J Biol Macromol. 2018 Dec;120(Pt B):1682-1695. doi: 10.1016/j.ijbiomac.2018.09.188. Epub 2018 Oct 1. PMID 30287361
- [Background] Callan P, Goodman GJ, Carlisle I, Liew S, Muzikants P, Scamp T, Halstead MB, Rogers JD. Efficacy and safety of a hyaluronic acid filler in subjects treated for correction of midface volume deficiency: a 24 month study. Clin Cosmet Investig Dermatol. 2013 Mar 20;6:81-9. doi: 10.2147/CCID.S40581. Print 2013. PMID 23687448
- [Background] Rippa AL, Kalabusheva EP, Vorotelyak EA. Regeneration of Dermis: Scarring and Cells Involved. Cells. 2019 Jun 18;8(6):607. doi: 10.3390/cells8060607. PMID 31216669
- [Background] Chen WY, Abatangelo G. Functions of hyaluronan in wound repair. Wound Repair Regen. 1999 Mar-Apr;7(2):79-89. doi: 10.1046/j.1524-475x.1999.00079.x. PMID 10231509
- [Background] De Boulle K, Heydenrych I. Patient factors influencing dermal filler complications: prevention, assessment, and treatment. Clin Cosmet Investig Dermatol. 2015 Apr 15;8:205-14. doi: 10.2147/CCID.S80446. eCollection 2015. PMID 25926750
- [Background] Dong J, Gantz M, Goldenberg G. Efficacy and safety of new dermal fillers. Cutis. 2016 Nov;98(5):309-313. PMID 28040813
- [Background] Draaijers LJ, Tempelman FR, Botman YA, Tuinebreijer WE, Middelkoop E, Kreis RW, van Zuijlen PP. The patient and observer scar assessment scale: a reliable and feasible tool for scar evaluation. Plast Reconstr Surg. 2004 Jun;113(7):1960-5; discussion 1966-7. doi: 10.1097/01.prs.0000122207.28773.56. PMID 15253184
- [Background] Eming SA, Martin P, Tomic-Canic M. Wound repair and regeneration: mechanisms, signaling, and translation. Sci Transl Med. 2014 Dec 3;6(265):265sr6. doi: 10.1126/scitranslmed.3009337. PMID 25473038
- [Background] Fakhari A, Berkland C. Applications and emerging trends of hyaluronic acid in tissue engineering, as a dermal filler and in osteoarthritis treatment. Acta Biomater. 2013 Jul;9(7):7081-92. doi: 10.1016/j.actbio.2013.03.005. Epub 2013 Mar 15. PMID 23507088
- [Background] Few J, Cox SE, Paradkar-Mitragotri D, Murphy DK. A Multicenter, Single-Blind Randomized, Controlled Study of a Volumizing Hyaluronic Acid Filler for Midface Volume Deficit: Patient-Reported Outcomes at 2 Years. Aesthet Surg J. 2015 Jul;35(5):589-99. doi: 10.1093/asj/sjv050. Epub 2015 May 11. PMID 25964628
- [Background] Fitzgerald R, Graivier MH, Kane M, Lorenc ZP, Vleggaar D, Werschler WP, Kenkel JM. Update on facial aging. Aesthet Surg J. 2010 Jul-Aug;30 Suppl:11S-24S. doi: 10.1177/1090820X10378696. PMID 20844296
- [Background] Freedberg et al. Fitzpatrick's Dermatology In General Medicine (Two Vol. Set) 6th edition (May 23, 2003
- [Background] Funt D, Pavicic T. Dermal fillers in aesthetics: an overview of adverse events and treatment approaches. Plast Surg Nurs. 2015 Jan-Mar;35(1):13-32. doi: 10.1097/PSN.0000000000000087. PMID 25730536
- [Background] Ghooi RB, Bhosale N, Wadhwani R, Divate P, Divate U. Assessment and classification of protocol deviations. Perspect Clin Res. 2016 Jul-Sep;7(3):132-6. doi: 10.4103/2229-3485.184817. PMID 27453830
- [Background] Grablowitz D, Ivezic-Schoenfeld Z, Federspiel IG, Gehl B, Kopera D, Prinz M. Long-term effectiveness of a hyaluronic acid soft tissue filler in patients with facial lipoatrophy, morphological asymmetry, or debilitating scars. J Cosmet Dermatol. 2020 Oct;19(10):2536-2541. doi: 10.1111/jocd.13454. Epub 2020 Jun 22. PMID 32333705
- [Background] Jiang LI, Stephens TJ, Goodman R. SWIRL, a clinically validated, objective, and quantitative method for facial wrinkle assessment. Skin Res Technol. 2013 Nov;19(4):492-8. doi: 10.1111/srt.12073. Epub 2013 Jun 10. PMID 23750828
- [Background] Kim BW, Moon IJ, Yun WJ, Chung BY, Kim SD, Lee GY, Chang SE. A Randomized, Evaluator-Blinded, Split-Face Comparison Study of the Efficacy and Safety of a Novel Mannitol Containing Monophasic Hyaluronic Acid Dermal Filler for the Treatment of Moderate to Severe Nasolabial Folds. Ann Dermatol. 2016 Jun;28(3):297-303. doi: 10.5021/ad.2016.28.3.297. Epub 2016 May 25. PMID 27274627
- [Background] Kim JH, Kwon TR, Lee SE, Jang YN, Han HS, Mun SK, Kim BJ. Comparative Evaluation of the Effectiveness of Novel Hyaluronic Acid-Polynucleotide Complex Dermal Filler. Sci Rep. 2020 Mar 20;10(1):5127. doi: 10.1038/s41598-020-61952-w. PMID 32198443
- [Background] Kopera D, Ivezic-Schoenfeld Z, Federspiel IG, Grablowitz D, Gehl B, Prinz M. Treatment of facial lipoatrophy, morphological asymmetry, or debilitating scars with the hyaluronic acid dermal filler Princess(R) FILLER. Clin Cosmet Investig Dermatol. 2018 Nov 27;11:621-628. doi: 10.2147/CCID.S181964. eCollection 2018. PMID 30568476
- [Background] Kopera D, Palatin M, Bartsch R, Bartsch K, O'Rourke M, Holler S, Baumgartner RR, Prinz M. An open-label uncontrolled, multicenter study for the evaluation of the efficacy and safety of the dermal filler Princess VOLUME in the treatment of nasolabial folds. Biomed Res Int. 2015;2015:195328. doi: 10.1155/2015/195328. Epub 2015 Mar 3. PMID 25821787
- [Background] Kuhne U, Esmann J, von Heimburg D, Imhof M, Weissenberger P, Sattler G. Safety and performance of cohesive polydensified matrix hyaluronic acid fillers with lidocaine in the clinical setting - an open-label, multicenter study. Clin Cosmet Investig Dermatol. 2016 Oct 20;9:373-381. doi: 10.2147/CCID.S115256. eCollection 2016. PMID 27799807
- [Background] Laurent TC, Fraser JR. Hyaluronan. FASEB J. 1992 Apr;6(7):2397-404. PMID 1563592
- [Background] Lemperle G, Holmes RE, Cohen SR, Lemperle SM. A classification of facial wrinkles. Plast Reconstr Surg. 2001 Nov;108(6):1735-50; discussion 1751-2. doi: 10.1097/00006534-200111000-00048. PMID 11711957
- [Background] Mashiko T, Kinoshita K, Kanayama K, Feng J, Yoshimura K. Perpendicular Strut Injection of Hyaluronic Acid Filler for Deep Wrinkles. Plast Reconstr Surg Glob Open. 2015 Dec 9;3(11):e567. doi: 10.1097/GOX.0000000000000552. eCollection 2015 Nov. PMID 26893992
- [Background] McCall-Perez F, Stephens TJ, Herndon JH Jr. Efficacy and tolerability of a facial serum for fine lines, wrinkles, and photodamaged skin. J Clin Aesthet Dermatol. 2011 Jul;4(7):51-4. PMID 21779421
- [Background] Park KY, Seok J, Rho NK, Kim BJ, Kim MN. Long-chain polynucleotide filler for skin rejuvenation: efficacy and complications in five patients. Dermatol Ther. 2016 Jan-Feb;29(1):37-40. doi: 10.1111/dth.12299. Epub 2015 Nov 2. PMID 26814448
- [Background] Poetschke J, Gauglitz GG. Current options for the treatment of pathological scarring. J Dtsch Dermatol Ges. 2016 May;14(5):467-77. doi: 10.1111/ddg.13027. PMID 27119465
- [Background] Rivkin AZ. Volume correction in the aging hand: role of dermal fillers. Clin Cosmet Investig Dermatol. 2016 Aug 30;9:225-32. doi: 10.2147/CCID.S92853. eCollection 2016. PMID 27621659
- [Background] Rumsey N. Psychosocial adjustment to skin conditions resulting in visible difference (disfigurement): What do we know? Why don't we know more? How shall we move forward? Int J Womens Dermatol. 2017 Dec 15;4(1):2-7. doi: 10.1016/j.ijwd.2017.09.005. eCollection 2018 Mar. PMID 29872669
- [Background] Rzany B, Cartier H, Kestemont P, Trevidic P, Sattler G, Kerrouche N, Dhuin JC, Ma YM. Full-face rejuvenation using a range of hyaluronic acid fillers: efficacy, safety, and patient satisfaction over 6 months. Dermatol Surg. 2012 Jul;38(7 Pt 2):1153-61. doi: 10.1111/j.1524-4725.2012.02470.x. PMID 22759252
- [Background] Savoia A., Onori N., Bladi A., Efficacy of Skinfill plus filler in the management of facial aging: a multicenter, post-marketing clinical study, Biomedical Dermatology volume 2, Article number: 2 (2018).
- [Background] Stephens TJ, Sigler ML, Herndon JH Jr, Dispensa L, Le Moigne A. A placebo-controlled, double-blind clinical trial to evaluate the efficacy of Imedeen((R)) Time Perfection((R)) for improving the appearance of photodamaged skin. Clin Cosmet Investig Dermatol. 2016 Mar 15;9:63-70. doi: 10.2147/CCID.S98787. eCollection 2016. PMID 27042135
- [Background] Sudha PN, Rose MH. Beneficial effects of hyaluronic acid. Adv Food Nutr Res. 2014;72:137-176. doi: 10.1016/B978-0-12-800269-8.00009-9. PMID 25081082
- [Background] van de Kar AL, Corion LU, Smeulders MJ, Draaijers LJ, van der Horst CM, van Zuijlen PP. Reliable and feasible evaluation of linear scars by the Patient and Observer Scar Assessment Scale. Plast Reconstr Surg. 2005 Aug;116(2):514-22. doi: 10.1097/01.prs.0000172982.43599.d6. PMID 16079683
- [Background] Van Dyke S, Hays GP, Caglia AE, Caglia M. Severe Acute Local Reactions to a Hyaluronic Acid-derived Dermal Filler. J Clin Aesthet Dermatol. 2010 May;3(5):32-5. PMID 20725567
- [Background] van Eijk T, Braun M. A novel method to inject hyaluronic acid: the Fern Pattern Technique. J Drugs Dermatol. 2007 Aug;6(8):805-8. PMID 17763611
- [Background] Zaleski-Larsen LA, Fabi SG, McGraw T, Taylor M. Acne Scar Treatment: A Multimodality Approach Tailored to Scar Type. Dermatol Surg. 2016 May;42 Suppl 2:S139-49. doi: 10.1097/DSS.0000000000000746. PMID 27128240